CLINICAL TRIAL: NCT07364682
Title: Assessment of Cardiac Function Using 2D Speckle Tracking Echocardiography (STE) in Neonates.
Brief Title: Measuring Heart Health in Both Term, Preterm and Unwell Newborn Babies With an Advanced Ultrasound Method: Speckle Tracking Echocardiography
Status: Not yet recruiting | Type: Observational
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Asad Abbas, Consultant Neonatologist, Birmingham Women's NHS Foundation Trust
Other Study IDs: 25/BW/OGN/NO/984
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Premature Baby; Pulmonary Hypertension of Newborn; Hypoxic Ischaemic Encephalopathy (HIE); Congenital Diaphragmatic Hernia; Chronic Lung DIsease
Keywords: Speckle Tracking Echocardiography; STE; Functional echocardiography; Neonatal Performed Echocardiography
MeSH Terms: conditions — Premature Birth; Hypoxia-Ischemia, Brain; Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Congenital Diaphragmatic Hernia: Term neonates diagnosed with Congenital Diaphragmatic Hernia (CDH)
- Hypoxic Ischaemic Encephalopathy: Term neonates diagnosed with Hypoxic Ischaemic Encephalopathy (HIE) and receiving therapeutic hypothermia.
- Acute pulmonary hypertension: Term neonates diagnosed with Acute Pulmonary Hypertension of the Newborn (aPHN), excluding those with CDH.
- Bronchopulmonary Dysplasia: Preterm neonates born at or before 32 weeks' gestation, who are later diagnosed with Chronic Lung Disease (CLD) requiring supplemental oxygen at 36 weeks corrected gestational age.
- Healthy preterms: (<36 weeks' gestation) admitted to the NICU and transitional care. Stratified into extreme preterm, moderately preterm and late preterm.
- Healthy term controls: (>36 weeks' gestation) who are well and on postnatal wards.

SUMMARY:
This study aims to improve how neonatologists check the heart function of newborn babies, especially those who are sick. While standard heart ultrasound scans are useful, a more advanced and sensitive technique called 2D speckle tracking echocardiography (STE) can detect subtle problems with how the heart muscle squeezes and relaxes. This may allow doctors to spot potential issues earlier.

Our research will take place at Birmingham Women's Hospital. The investigators will perform these advanced, non-invasive heart scans on several groups of babies:

1. Healthy term and premature babies, to establish a "normal" range of heart function.
2. Babies who are unwell with specific conditions, including those with brain injury due to lack of oxygen at birth (HIE), chronic lung disease of prematurity (BPD), a hole in the diaphragm (CDH), or high blood pressure in their lungs (aPHN).

The heart scan is a standard, painless procedure. Using STE does not require any extra scanning time or cause any additional discomfort to the baby; the special images are taken during the routine scan. For many of the sick babies, these scans are already part of their normal clinical care.

The main goals of this observational study are to see if STE is a feasible and reliable tool in newborns, to establish normal values for healthy babies, and to track how heart function changes in sick babies during their illness and recovery.

Ultimately, the investigators hope this research will provide doctors with a better tool to assess heart health in newborns. This could lead to earlier, more accurate detection of heart problems and help guide treatment decisions to improve outcomes for these vulnerable infants.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who are inpatient at the Birmingham Women's Hospital
* Confirmed diagnosis of acute pulmonary hypertension, congenital diaphragmatic hernia, hypoxic ischaemic encephalopathy, or bronchopulmonary dysplasia/chronic lung disease (defined by oxygen/respiratory support requirement at 36 weeks post menstrual/corrected gestational age).

OR

* Health control (>36 weeks - well and on the postnatal ward)
* Well preterm neonate (<36 weeks) admitted to the NICU, transitional care or post-natal wards.
* Informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

* Presence of major congenital heart disease (other than patent foramen ovale or patent ductus arteriosus).
* Presence of other life-limiting congenital anomalies (other than CDH) or syndromes that could independently affect cardiac function.
* Inability to obtain adequate echocardiographic images for STE analysis after reasonable attempts.
* If the neonatal consultant or neonatal nurse caring for the neonate feels that the neonate is too unstable for inclusion in the study or that consent should not be sought from parents.

Ages: 0 Minutes to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Inpatient status at Birmingham Women's Hospital Neonatal Unit - only babies admitted to the neonatal unit, transitional care ward or postnatal ward will be considered for screening.
  Belong to one of the following target clinical groups:
  * Group 1: Term neonates diagnosed with Hypoxic Ischaemic Encephalopathy (HIE) and receiving therapeutic hypothermia.
  * Group 2: Preterm neonates born at or before 32 weeks' gestation, who are later diagnosed with Chronic Lung Disease (CLD) requiring supplemental oxygen at 36 weeks corrected gestational age.
  * Group 3: Term neonates diagnosed with Congenital Diaphragmatic Hernia (CDH).
  * Group 4: Term neonates diagnosed with Acute Pulmonary Hypertension of the Newborn (aPHN), excluding those with CDH.
  * Healthy controls:
  * Term neonates (>36 weeks' gestation) who are well and on postnatal wards.
  * Well preterm neonates (<36 weeks' gestation). • Stable enough for echocardiography and research inclusion, as determined by the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of acquiring adequate quality images for comprehensive Right ventricular - Speckle Tracking Echocardiography (RV-STE), Left ventricular (LV) STE, and left atrial (LA) -STE in neonates with aPHN, CDH, HIE, and BPD. | By completion of data collection (September 2027)
  Feasibility rate of RV, LV, and LA STE.
To describe the longitudinal changes in RV, LV, and LA STE parameters from acute illness through recovery/discharge in each disease cohort. | By September 2027
  The invetigators will measure this by looking at values and longitudinal trends of: RV-Global Longitudinal Strain (GLS), RV-Free Wall Longitudinal Strain (FWLS), LV-GLS, LA reservoir strain (LASr) in healthy neonates and neonates with disease conditions (HIE, BPD, CDH, aPHN).
To establish normative values of simultaneously performed RV, LV and LA strain in well term and preterm neonates | By September 2027
  The investigators will establish normative reference RV, LV and LA strain using two-dimensional speckle-tracking echocardiography in a cohort of well term and preterm neonates. Report Strain values as means ± standard deviations and percentiles (5th-95th), stratified by gestational age, postnatal age, and birth weight categories.

SECONDARY OUTCOMES:
To evaluate the intra-observer and inter-observer reproducibility of RV, LV, and LA STE measurements | By September 2027
  The investigators will use intra-class correlation coefficients (ICC), Bland-Altman limits of agreement, and coefficient of variation (CV) for key STE parameters.
To compare STE-derived parameters with conventional echocardiographic measures of cardiac function. | By September 2027
  Correlation and agreement between speckle tracking echocardiography (STE)-derived parameters (STE derived EF, STE derived TAPSE) and conventional echocardiographic measures of cardiac function (EF by Simpson Biplane technique, M-mode TAPSE).
To compare RV, LV, and LA STE parameters between the different disease cohorts and a cohort of healthy control neonate | By September 2027
  Comparison of right ventricular (RV), left ventricular (LV), and left atrial (LA) strain and strain rate parameters derived from speckle tracking echocardiography (STE) between neonates in different disease cohorts and a healthy control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham Women's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial will be available upon reasonable request to the CI.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The study protocol will be published as part of registration on clinicaltrials.gov.
  The anonymised participant-level dataset, statistical code, and Final Study Report may be made available through institutional repositories or by request, subject to ethical approvals, consent, and data protection safeguards.
  These materials will be shared no later than 12 months after final study reporting or publication.
  Access will require appropriate agreements and will follow national guidance on open data sharing.
Access Criteria: De-identified individual participant data (IPD) from this study will be available upon reasonable request to the Chief Investigator, subject to approval of a study proposal and any necessary data-sharing agreements.